CLINICAL TRIAL: NCT02760212
Title: Physical Approaches to the Management of Fibromyalgia - A Multidisciplinary Approach
Brief Title: Treatment and Assessment of Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lakehead University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LakeheadU
Record Dates: First submitted 2016-04-20; First posted 2016-05-03 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Fibromyalgia
Keywords: Shockwave therapy; fMRI; blood biomarkers
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Radial Shockwave Therapy Group (Experimental): Participants in Group 1 will receive RSWT to the most painful spot within each of the 3 most painful regions as described by the participant. Treatments will be spaced one week apart over a 5 week period of time. 5 weekly sessions with treatment to the painful areas will be undertaken with 500 shocks (1.5 bar, 15 Hz), then 1000 shocks (2 bar, 8 Hz), and finally 500 shocks (1.5 bar, 15 Hz) to the most painful spot.
  Interventions: Device: Radial Shockwave Therapy
- Group 2 - Placebo Group (Placebo Comparator): Participants in Group 2 will receive a placebo treatment with a soft rubber cap applied to the applicator, leaving air between the transmitter and the cap and the participant's skin so that no shockwave will be generated nor applied to the participant's skin. Treatments will be spaced one week apart over a 5 week period of time. 5 weekly sessions with placebo treatment to the painful areas will be undertaken with 2000 placebo shocks (15 Hz) producing an audible sound but no therapeutic dosage to the most painful spot. Upon completion of the placebo treatment, participant's will be offered the experimental treatment but this data will not be used for comparison and analysis.
  Interventions: Other: Placebo Comparator: Group 2 - Placebo Group

INTERVENTIONS:
Device: Radial Shockwave Therapy — 5 treatments in total scheduled weekly; RSWT to the painful areas will be undertaken with 500 shocks (1.5 bar, 15 Hz), then 1000 shocks (2 bar, 8 Hz), and finally 500 shocks (1.5 bar, 15 Hz) to the most painful spot within each of the 3 most painful regions as described by the participant.
  Other Names: Storz D-Actor 100
  Arms: Group 1 - Radial Shockwave Therapy Group
Other: Placebo Comparator: Group 2 - Placebo Group — 5 treatments in total scheduled weekly; placebo to the painful areas will be undertaken with 2000 shocks to the most painful spot within each of the 3 most painful regions as described by the participant.
  Other Names: Storz D-Actor 100
  Arms: Group 2 - Placebo Group

SUMMARY:
Fibromyalgia is a common disorder affecting approximately 2% of the Canadian population. Patients diagnosed with fibromyalgia commonly present with chronic, widespread pain as well as fatigue, depression, mood disturbances, and cognitive symptoms. As a result, fibromyalgia has a negative impact on the patient's quality of life, and a negative financial impact for them, society, and the healthcare system, through lost wages and delayed diagnosis. Therefore a more direct and conclusive method of diagnosis is needed.

Recently, fibromyalgia diagnosis has been based on the modified American College of Rheumatology Preliminary Diagnostic Criteria for fibromyalgia. To assist with diagnosis, recent evidence shows that compared to healthy people, people with fibromyalgia present with differences on functional MRI (fMRI) whole brain scans, as well as differences in a functional blood biomarker challenge test, known as fm/a. The fm/a determines the function of the immune system in response to a stimulus, and has been used previously to show that people with fibromyalgia have a severely blunted immune response.

Despite the number of treatment options available, interventions for chronic pain remain largely ineffective. In light of its demonstrated effectiveness, safety, and ease of use in previous studies, radial shockwave therapy (RSWT) has been selected for inclusion in the present study. The main objective of this study is to determine the efficacy and effect of RSWT compared to placebo on the symptoms frequently reported in association with fibromyalgia. In addition, the fm/a and brain activity associated with pain patterns (fMRI) may assist in early diagnosis and prediction of treatment success in patients with fibromyalgia.

DETAILED DESCRIPTION:
At St. Joseph's Care Group (SJCG) rheumatologist and chronic pain physician will determine if a client is eligible to participate in the study using the inclusion/exclusion criteria (outlined in the attached grant proposal). Physician would then ask if the client would be open to discussing their possible involvement in a research study. If so, a member of the research team other than physicians will visit with the client at the Chronic Pain Management program at SJCG to discuss the project and complete the informed consent process if the client would like to participate.

Following informed consent, the participant would be assigned to one of two groups following a restricted randomization procedure. This will be completed using open-source minimization software called Qminim. The process of minimization ensures group sizes are equal and eliminates potential bias that may be introduced which is important for clinical research of small sizes. Group 1 will receive Radial Shockwave Therapy (RSWT) while group 2 will be the placebo group. Once participants in the placebo group have completed the study, RSWT will be offered, although it will not be included in the data analysis. Participants will be grouped for minimization based on sex and age in the following ranges: 18-30, 31-45, 46-60 years. All participant information/group assignment will be coded to maintain confidentiality. Group assignment will be unknown to the participant until they complete the study (or withdraw from the study).

The following initial assessments will occur prior to receiving the RSWT or placebo: At SJCG: participants will undergo quantitative sensory testing for allodynia and hyperalgesia by one of the physicians. At Lakehead University School of Kinesiology: participants will have basic demographic information such as height, weight and age, measured and recorded on a data abstraction form by a member of the research team. The participant will also be asked to consider the most painful spot within each of the 3 most painful regions in his/her body. Participants will mark on a 100 millimeter VAS scale at the point that corresponds to the pain intensity for each region. The amount of pain will be estimated by measuring in millimeters the distance from the "no pain" marker to the mark provided by the participant for each question. This will be recorded on the data abstraction form. Pressure pain threshold will next be measured on the most painful spot within each of the 3 most painful regions using a Baseline© Pressure Tolerance Meter (60 lbs). Pressure will be applied perpendicular to the tissue in the three most painful regions as indicated by the participant. The participant will be asked to report when the pressure applied to the region became painful and the amount of pressure shall be recorded in pounds on the data abstraction form. A 30 second rest shall be allowed for recovery and the same technique shall be applied to the other painful locations. The specific location of the painful region shall be marked and documented by a trained member of the research team. Next, participants will be asked to complete the Beighton Scoring Screen for hypermobility, Beck's Depression Scale, and Pain Catastrophizing Scale questionnaires. All scores will be recorded on the data abstraction form. At Lakehead University (NOSM rooms 1002A, C, D E, F or School of Kinesiology SB-1028): participants will be scheduled to have a blood sample drawn by a registered phlebotomist. Specialized vacutainers will be used to isolate Peripheral Blood Mononuclear Cells (PBMCs) which will be later used in cytokine protein analysis. All blood taken will be labeled with a participant code to maintain confidentiality, and stored at NOSM.

At TBRHSC: 15 randomly selected participants from each group will undergo whole brain functional MRI (fMRI) imaging by a member of the research team at TBRHSC. The scans will include a resting state fMRI, an 8 minute scan during alternating 30 second on, 30 second off evoked pressure pain stimulus, a T1 high resolution anatomical image, and a diffusion tensor image. Please see the attached grant proposal for details regarding this imaging method.

Once the initial measures are completed, participants will be scheduled to begin the allocated treatment based on group assignment. Group 1 will receive RSWT to the most painful spot within each of the 3 most painful regions, while group 2 (placebo) will receive a similar treatment but a soft rubber cap will be applied to the applicator, leaving air between the transmitter and the cap and the participant's skin. Treatments will be spaced one week apart over a 5 week period of time and will occur at Lakehead University's School of Kinesiology, room SB-1028.

Upon completion of the treatments, participants will complete the same measures/questionnaires that were performed at the beginning of the study. Also, one vial of blood will be taken again and if the participant was in the fMRI group, they will repeat the same imaging sessions detailed above.

At the conclusion of the study, participants will be invited to participate in a focus group lead by another research team member during which qualitative feedback regarding the study will be discussed. This is a patient-centred approach that will help the investigators engage the fibromyalgia community and allow this input to guide future study design.

It is anticipated that 50 participants will be enrolled in the study. The main analysis will be a comparison of the pre- and post-outcomes, meaning that this is a repeated measures study design. This design has the advantage of minimizing the effect of inter-subject variability. A power analysis was performed a priori and it was determined that this sample size is sufficient; minimum detectable differences of 10% and standard deviation of ±15% resulting in a power of 0.892.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-60 years
2. diagnosed with FM by a physician based on ARC Diagnostic Criteria\
3. willing to provide informed consent to be randomized to either of the treatment pathways and willing to follow the study protocol
4. have no contraindications to MRI (determined by MRI safety screening with a licensed MRI technologist).

Exclusion Criteria:

1. Have any vascular, neurological, or other condition or disorder (e.g., rheumatoid arthritis, osteoarthritis) that could reasonably explain pain
2. have implanted metal non compatible with MRI or shockwave therapy
3. are pregnant
4. are diagnosed with thrombosis, thrombophlebitis, or coagulation disorders
5. have anxiety or claustrophobia that will be aggravated by the confined spaces of the fMRI.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) Pain Score from Baseline to 6 Weeks | Measured pre-treatment (baseline) and post-treatment (at 6 weeks)
  Subject pain will be rated using a VAS by the participant for the 3 most painful regions.

SECONDARY OUTCOMES:
Focus Group Qualitative Themes Identified from Transcripted Survey Responses | Post-treatment (at 6 weeks)
  Participants will be invited to participate in a focus group lead by a member of the research team during which qualitative feedback regarding the study will be discussed. This is a patient-centred approach that will help the investigators engage the fibromyalgia community and allow this input to guide future study design.
Change in Pressure Pain Threshold from Baseline to 6 Weeks | Measured pre-treatment (baseline) and post-treatment (at 6 weeks)
  Pressure pain threshold will be measured on the most painful spot within each of the 3 most painful regions using a Baseline© Pressure Tolerance Meter (60 lbs). Pressure will be applied perpendicular to the tissue in the 3 most painful regions as indicated by the participant. The participant will be asked to report when the pressure applied to the region became painful and the amount of pressure shall be recorded in pounds on the data abstraction form. A 30 second rest shall be allowed for recovery and the same technique shall be applied to the other painful locations. The specific location of the painful region shall be marked and documented by a trained member of the research team.
Change in Blood Biomarker fMA Test from Baseline to 6 Weeks | Measured pre-treatment (baseline) and post-treatment (at 6 weeks)
  A blood sample will be drawn by a registered phlebotomist. Specialized vacutainers will be used to isolate Peripheral Blood Mononuclear Cells (PBMCs) which will be later used in cytokine protein analysis.
Change in Functional Magnetic Resonance Imaging from Baseline to 6 Weeks | Measured pre-treatment (baseline) and post-treatment (at 6 weeks)
  Resting State fMRI - An 8 minute task free scan will be acquired to investigate alterations in the functional connectivity of the default mode network, found previously to be altered in chronic pain conditions including FM. Recruitment of the pain matrix - An 8 minute scan with an alternating 30 second on and 30 second off evoked pressure pain stimulus applied to the affected area. T1 high resolution anatomical imaging - This scan lasting about 8 minutes is used for the registration of functional images to allow group fMRI analysis as well as for overlay purposes. It will also be used to evaluate grey matter volume through a VBM analysis. Diffusion Tensor Image - This 9 minute scan allows visualization of the white matter tracts and will be used for evaluation of white matter integrity.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Sanzo, DScPT, Principal Investigator — Lakehead University
Locations (1):
- Lakehead University, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Potential participants will have the opportunity to indicate that they would like individual results of study and provide contact information so that contact can be made upon completion of the study and information can be provided at that time.
Supporting Information: CSR
Time Frame: Study participants may obtain a summary report of the study results upon completion of analysis and publication of findings.
Access Criteria: Study participants may contact research team for information.
URL: https://tbay.research@gmail.com

REFERENCES:
- [Derived] Sanzo P, Agostino M, Fidler W, Lawrence-Dewar J, Pearson E, Zerpa C, Niccoli S, Lees SJ. Shockwave therapy and fibromyalgia and its effect on pain, blood markers, imaging, and participant experience - a multidisciplinary randomized controlled trial. Physiother Theory Pract. 2025 Jan;41(1):99-114. doi: 10.1080/09593985.2024.2321503. Epub 2024 Feb 21. PMID 38384123